CLINICAL TRIAL: NCT00920959
Title: A Stratified, Randomized, Double-blind, Placebo-controlled, Parallel-group, 12 Week Trial Evaluating the Safety and Efficacy of Fluticasone Propionate/Salmeterol DISKUS Combination Product 100/50mcg Once Daily Versus Fluticasone Propionate DISKUS 100mcg Once Daily and Placebo in Symptomatic Pediatric Subjects (4-11 Years) With Asthma
Brief Title: Advair Pediatric Once-Daily
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SAS30021
Record Dates: First submitted 2009-06-12; First posted 2009-06-15 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Fluticasone propionate/salmeterol combination (Experimental): study drug
  Interventions: Drug: FSC 100/50mcg
- Fluticasone propionate (Experimental): study drug
  Interventions: Drug: FP 100mcg
- Placebo (Experimental): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FP 100mcg — Once-daily dosing
  Arms: Fluticasone propionate
Drug: FSC 100/50mcg — Once-daily dosing
  Arms: Fluticasone propionate/salmeterol combination
Drug: Placebo — Once-daily dosing
  Arms: Placebo

SUMMARY:
To demonstrate if once-daily dosing of ADVAIR 100/50 once-daily has superior efficacy and comparable safety compared with FP 100mcg once-daily in pediatric subjects 4 to 11 years of age with asthma.

ELIGIBILITY:
Inclusion Criteria:

* Out-patients
* Asthma diagnosis
* Reversibility
* Short-acting beta-agonist or asthma controlled medication use

Exclusion Criteria:

* Life-threatening asthma
* Specified asthma medications
* Chickenpox
* Drug allergy
* Respiratory infections
* Tobacco use
* Clinical laboratory abnormalities
* Ophthalmologic conditions
* Investigation medications
* Affiliation with investigator site

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 908 (Actual)
Dates: Start 2001-11; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline at endpoint in daily PM PEF | 12 weeks

SECONDARY OUTCOMES:
Various pulmonary function endpoints | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (129):
- United States (121):
  - GSK Investigational Site, Ozark, Alabama
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Crescent City, California
  - GSK Investigational Site, Dinuba, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, La Jolla, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Mission Viejo, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Orange, California
  - GSK Investigational Site, Palmdale, California
  - GSK Investigational Site, Panorama City, California
  - GSK Investigational Site, Paramount, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Rolling Hills Estates, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, San Jose, California
  - GSK Investigational Site, Sherman Oaks, California
  - GSK Investigational Site, Vista, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Centennial, Colorado
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Pueblo, Colorado
  - GSK Investigational Site, Altamonte Springs, Florida
  - GSK Investigational Site, Hialeah, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Tallahassee, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Barnesville, Georgia
  - GSK Investigational Site, Martinez, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Glenview, Illinois
  - GSK Investigational Site, Hoffman Estates, Illinois
  - GSK Investigational Site, Park Ridge, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, South Bend, Indiana
  - GSK Investigational Site, Lawrence, Kansas
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Murray, Kentucky
  - GSK Investigational Site, Covington, Louisiana
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Sunset, Louisiana
  - GSK Investigational Site, Newton, Massachusetts
  - GSK Investigational Site, North Dartmouth, Massachusetts
  - GSK Investigational Site, Taunton, Massachusetts
  - GSK Investigational Site, West Quincy, Massachusetts
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Columbia, Missouri
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Missoula, Montana
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Papillion, Nebraska
  - GSK Investigational Site, Berlin, New Jersey
  - GSK Investigational Site, Brick, New Jersey
  - GSK Investigational Site, East Orange, New Jersey
  - GSK Investigational Site, Ocean City, New Jersey
  - GSK Investigational Site, Verona, New Jersey
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, Liverpool, New York
  - GSK Investigational Site, New Hyde Park, New York
  - GSK Investigational Site, Rockville Centre, New York
  - GSK Investigational Site, Vestal, New York
  - GSK Investigational Site, Asheville, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Elizabeth City, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Bend, Oregon
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Altoona, Pennsylvania
  - GSK Investigational Site, Blue Belle, Pennsylvania
  - GSK Investigational Site, Harrisburg, Pennsylvania
  - GSK Investigational Site, Lewisburg, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Upland, Pennsylvania
  - GSK Investigational Site, Lincoln, Rhode Island
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Mt. Pleasant, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, El Paso, Texas
  - GSK Investigational Site, Galveston, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Lake Jackson, Texas
  - GSK Investigational Site, New Braunfels, Texas
  - GSK Investigational Site, Plano, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Layton, Utah
  - GSK Investigational Site, Murray, Utah
  - GSK Investigational Site, Burke, Virginia
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Edmonds, Washington
  - GSK Investigational Site, Tacoma, Washington
  - GSK Investigational Site, Charleston, West Virginia
  - GSK Investigational Site, Greenfield, Wisconsin
  - GSK Investigational Site, La Crosse, Wisconsin
- Argentina (3):
  - GSK Investigational Site, Buenos Aires, Buenos Aires
  - GSK Investigational Site, Santa Fe, Santa Fe Province
  - GSK Investigational Site, Buenos Aires
- Chile (2):
  - GSK Investigational Site, Viña del Mar, Región de Valparaíso
  - GSK Investigational Site, Santiago, Región Metro de Santiago
- GSK Investigational Site, Breña, Peru
- Puerto Rico (2):
  - GSK Investigational Site, Ponce, Puerto Rico
  - GSK Investigational Site, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] This study has not been published in the scientific literature.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: SAS30021 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: SAS30021 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: SAS30021 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: SAS30021 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: SAS30021 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: SAS30021 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: SAS30021 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register